CLINICAL TRIAL: NCT07279142
Title: Efficacy and Safety of 7 Millimeters Vaginal Radiofrequency in Overactive Bladder
Acronym: HYPNOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Università della Campania Luigi Vanvitelli (Unknown)
Responsible Party: Principal Investigator, Stefano Salvatore, Professor, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYPNOS
Record Dates: First submitted 2025-11-19; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Overactive Bladder (OAB); Incontinence, Urge
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients who have never received pharmacological or medical device treatment for OAB (Experimental): Transvaginal micro-radiofrequency with 7mm needles in patients who have never received pharmacological or medical device treatment for OAB (first-line group).
  Interventions: Device: Radiofrequency
- patients who have failed adequate therapy (≥12 weeks) with antimuscarinics (Experimental): Transvaginal micro-radiofrequency with 7 mm needles in patients who have failed adequate therapy (≥12 weeks) with antimuscarinics due to ineffectiveness, intolerance or contraindications (refractory group)
  Interventions: Device: Radiofrequency

INTERVENTIONS:
Device: Radiofrequency — According to the study protocol, eligible subjects will receive one treatment within 3 weeks of screening. After one month, if there is no satisfactory result, a second treatment will be administered, and after another month, the patient will be evaluated. If there is still no end point, a third treatment will be given. It should be noted that the second and third treatments will only be performed if there is no satisfactory result after the previous treatment. Treatment area: Treatment area will include vaginal canal.
  Treatment Procedure:
  * Subjects receive HYPNOS treatment with device using radiofrequency (RF). Treat vaginal canal at the depth starting from approximately 3.5cm from introitus to the distal end of vagina. Radially the treatment area is from 9 to 3 o'clock.
  * Patient should empty bladder prior to treatment
  * Position patient in lithotomy position
  * Set energy to levels well tolerated by the subject. Suggested settings: Burst Mode 7mm, 1 pass.

SUMMARY:
The investigator hypothesizes that controlled delivery of low heat (45-50 Centigrade) to the sub-detrusor and detrusor muscle can ablate the autonomic nerve endings and control overactive bladder symptoms without causing significant damage to the surrounding structures. Low heat in such a manner is below urethral sensation and enables office treatment. The transvaginal approach is non-invasive and improves overactive bladder (OAB) symptoms and patients' quality of life. The investigator believes that the RF administration results could be equal or better for first-line treated patients compared to pharmacological refractory patients.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old
* Subject is willing to provide Informed Consent, is geographically stable, understands the requirements for completing the bladder diary and is willing to comply with the required diary, follow-up visits, and testing schedules.
* Urinary incontinence, predominant urgency incontinence, with moderate-severe overactive bladder, International Consultation on Incontinence Questionnaire - Overactibe Bladder Short Form (ICIQ-OABSS) score ≥6.
* Ability and willingness to self-catheterize in case this is necessary.
* With respect to their reproductive capacity must be post-menopausal or surgically sterile or willing to use a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly from screening until the last follow up

Exclusion Criteria:

* Pacemaker or internal defibrillator, or any other metallic or electronic implant anywhere in the body.
* Any permanent implant or an injected chemical substance in the treatment area.
* Superficial areas that have been injected with hyaluronic acid (HA)/collagen/fat injections or other augmentation methods with bio-material during last 6 months.
* Current or history of cancer, or current condition of any other type of cancer, or premalignant moles.
* Severe concurrent conditions, such as cardiac disorders, sensory disturbances, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy, the intention of pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as Acquired Immunodeficency Syndrome (AIDS) and Human Immunodeficency Virus (HIV), autoimmune disorders, or use of immunosuppressive medications.
* Patients with a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction and hormonal virilization.
* Any active condition in the treatment area, such as sores, eczema, and rash.
* History of vaginal disorders, keloids, abnormal wound healing.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days, as per the practitioner's discretion.
* Non-italian speakers
* Severely impaired mobility or cognition
* Spinal cord injury or advanced/severe neurologic condition including Multiple Sclerosis, Parkinson's Disease
* Repair of pelvic organ prolapse or incontinence procedure in the previous 6 months
* Ongoing complications of prior anti-incontinence surgery
* Received intravesical botulinum injection within the previous 12 months
* History of an implanted nerve stimulator for incontinence
* History of prior sling or vaginal mesh placement,
* Previous diagnosis of interstitial cystitis, bladder cancer, or chronic pelvic pain
* Current participation in any other conflicting interventional or OAB treatment study
* Planning to become pregnant during the study period.
* Pelvic radiation, history of pelvic radiation
* Active urinary tract or vaginal infection
* Anatomical conditions that would prevent the introduction and use of the device, in such as significant pelvic organ prolapse,
* Current hydronephrosis or hydroureter
* Bladder outflow obstruction
* Active pelvic organ malignancy
* Urethral obstruction
* Urinary retention or prolonged catheter use
* Less than 12 months post-partum or currently pregnant or plan to become pregnant in the following 12 months.
* Untreated symptomatic urinary tract infection
* Unevaluated hematuria
* Medical instability
* Allergy to anesthetics as Benzocaine/Lidocaine/Tetracaine Cream (BLT Cream) used in the study
* Not available for follow-up in 6 months
* Participation in other research trials that could influence results of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — With respect to their reproductive capacity must be post-menopausal or surgically sterile or willing to use a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly from screening until the last follow up
Enrollment: 48 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-11-13 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Improvement of 40% in the Overactive Bladder Symptoms Bother Questionnaire Score Short Form from the baseline score | From enrollment to 12 weeks after last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rovner ES, Versi E, Le Mai T, Dmochowski RR, De Wachter S. One-year results with selective bladder denervation in women with refractory overactive bladder. Neurourol Urodyn. 2019 Nov;38(8):2178-2184. doi: 10.1002/nau.24110. Epub 2019 Jul 29. PMID 31359508
- [Background] Abdelaziz A, Dell J, Karram M. Transvaginal radiofrequency energy for the treatment of urinary stress incontinence: A comparison of monopolar and bipolar technologies in both pre- and post-menopausal patients. Neurourol Urodyn. 2021 Sep;40(7):1804-1810. doi: 10.1002/nau.24748. Epub 2021 Jul 20. PMID 34288106
- [Background] Cespedes RD, Cross CA, McGuire EJ. Modified Ingelman-Sundberg bladder denervation procedure for intractable urge incontinence. J Urol. 1996 Nov;156(5):1744-7. PMID 8863585
- [Background] Dayan E, Ramirez H, Westfall L, Theodorou S. Role of Radiofrequency (Votiva, InMode) in Pelvic Floor Restoration. Plast Reconstr Surg Glob Open. 2019 Apr 25;7(4):e2203. doi: 10.1097/GOX.0000000000002203. eCollection 2019 Apr. PMID 31321190
- [Background] Takahashi T, Garcia-Osogobio S, Valdovinos MA, Belmonte C, Barreto C, Velasco L. Extended two-year results of radio-frequency energy delivery for the treatment of fecal incontinence (the Secca procedure). Dis Colon Rectum. 2003 Jun;46(6):711-5. doi: 10.1007/s10350-004-6644-8. PMID 12794570